CLINICAL TRIAL: NCT07134517
Title: Examining the Effects of Reformer Pilates Exercises on Physical Fitness and Cognitive Functions in Healthy Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, BÜŞRA CANDİRİ, Assistant Professor, Inonu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/8028
Record Dates: First submitted 2025-07-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers (HV)
Keywords: Pilates; cognitive function; physical fitness
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group in this study will consist of individuals who perform reformer Pilates exercises twice a week for a total of 16 sessions over an 8-week period.
  Interventions: Other: Pilates exercise
- Control group (No Intervention): The control group will consist of individuals who do not actively participate in reformer Pilates or any other sports activities.

INTERVENTIONS:
Other: Pilates exercise — The principles of centering, concentration, breathing, control, flow, and precision in the Pilates method will be explained to participants. Pelvic floor activity and lateral breathing will be taught and practiced, along with neutral spine alignment. The first and last 5 minutes of each session will consist of stretching exercises. Stretching exercises will begin with 3-5 repetitions, while strengthening and stabilization exercises will start with 6-8 repetitions, with the number of repetitions increasing each week based on participants' tolerance. Springs are attached according to the purpose and difficulty level of the exercises. Stretching exercises are performed with lighter resistance springs, while strengthening and stabilization exercises are performed with higher resistance springs. All movements will be demonstrated and explained to ensure the exercises are performed correctly. Verbal cues will be given for breath control and centering.
  Arms: Intervention group

SUMMARY:
Pilates is an exercise method that aims to increase body awareness and improve physical fitness through controlled movements based on mind-body integration. Reformer Pilates strengthens the mind-body connection while increasing core muscle activation through equipment-assisted exercises. It is known that regular exercise has positive effects on cognitive functions through its neuroprotective and neuroplastic effects. However, the effects of Reformer Pilates on these functions have been studied in only a limited number of studies, particularly in healthy middle-aged individuals. The aim of this project proposal is to investigate the effectiveness of Reformer Pilates exercises on physical fitness and cognitive functions in healthy individuals. In this study, the effects of reformer Pilates on physical fitness and cognitive functions will be examined in healthy individuals aged 18-50. The intervention group will perform reformer Pilates twice a week for 8 weeks, while the control group will not participate in any physical activity. Body mass index, waist-to-height ratio, waist-to-hip ratio, cognitive reserve, cognitive functions, reaction time, physical fitness, grip strength, and general health status will be assessed at baseline and after 8 weeks. Cognitive functions will be assessed using the cognitive reserve index, and cognitive functions will be assessed using the Stroop test-anchor form and the tracking test. Stroop test-anchor form and tracking test; reaction time will be measured using a wireless system consisting of a laser LED light emitter and a central hand control unit; physical fitness will be assessed using The Senior Fitness Test; grip strength will be measured using a hand dynamometer; and general health status will be assessed using the General Health Questionnaire-12. Data analysis will be performed using SPSS version 25.0. For comparing pre- and post-treatment outcome measures within the group, analysis will be conducted using the t-test for dependent samples (if normally distributed) or the Wilcoxon signed-rank test (if not normally distributed). Effect size will be calculated to determine the impact of the exercise program. P<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who do not have a regular exercise habit,
* Are between the ages of 18 and 50,
* And are inactive according to the International Physical Activity Questionnaire Short Form assessment (less than 600 MET min).

Exclusion Criteria:

* Individuals with a history of serious musculoskeletal or neurological disease,
* Receiving psychological support,
* Taking regular medication,
* With metabolic disease,
* Describing chronic pain anywhere in their body,
* Or with communication problems.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Stroop Test - Anchor Form | 8 weeks
  The Stroop Test, developed by Stroop in 1935, is a test used to assess selective attention, cognitive flexibility, inhibition skills, and information processing speed. Successful performance requires suppressing processes unrelated to the task and focusing on processes related to the task. There are many types of forms used in the Stroop Test. In Turkey, the Stroop Test Çapa form, whose validity and reliability were established by Emek Savaş et al., is widely used. In this study, the Stroop Test-Çapa Form will be used to assess individuals' cognitive flexibility. The test consists of a total of 60 items. A long test duration and a high number of errors indicate weak cognitive flexibility.

SECONDARY OUTCOMES:
Tracking test | 8 weeks
  It was developed by Reitan (1955). It measures executive functions such as working memory, complex attention, planning, and set-shifting abilities. It consists of two sections, A and B. Section A contains circles with numbers scattered on an A4 sheet of paper. In section A, participants are asked to connect the numbers inside the circles in order (1-2-3-...) by drawing a line. In section B, there are circles scattered on an A4 sheet of paper, but these circles contain both numbers and letters. In this section, participants are asked to connect the numbers and letters inside the circles in alternating order (1-A-2-B-...), one number followed by one letter. Section A assesses processing speed, while Section B assesses set-shifting, response inhibition, and interference resistance skills.
Reaction time (Time) | 8 weeks
  Upper and lower extremity reaction time will be measured using a wireless system consisting of a laser LED light emitter and a central hand control unit. For the lower extremity reaction time assessment, individuals are asked to extinguish four randomly lit LEDs placed on the ground at 1-meter intervals as quickly as possible within a 30-second time frame while standing on one foot. The assessment will be recorded separately for the right and left legs. The unit extinguishing time in milliseconds are recorded. For the upper extremity reaction time assessment, participants are asked to extinguish five LEDs on a table as quickly as possible with one hand while in a sitting position. The right and left hands are evaluated separately. The unit extinguishing time in milliseconds are recorded.
Reaction time (Count) | 8 weeks
  Upper and lower extremity reaction time will be measured using a wireless system consisting of a laser LED light emitter and a central hand control unit. For the lower extremity reaction time assessment, individuals are asked to extinguish four randomly lit LEDs placed on the ground at 1-meter intervals as quickly as possible within a 30-second time frame while standing on one foot. The assessment will be recorded separately for the right and left legs. The number of LEDs that can be extinguished within 30 seconds,and the number of LEDs missed after the 5-second light emission period are recorded. For the upper extremity reaction time assessment, participants are asked to extinguish five LEDs on a table as quickly as possible with one hand while in a sitting position. The right and left hands are evaluated separately.
Assessment of Physical Fitness | 8 weeks
  The Senior Fitness Test will be used to assess physical fitness. It consists of six functional tests that measure strength, endurance, balance, agility, and flexibility.
Grip Strength Test | 8 weeks
  Hand grip strength will be measured using a hand dynamometer. Participants will sit with their shoulders adducted alongside their torso, elbows flexed at 90°, forearms in a neutral position, and wrists in 0-30° extension and 0-15° ulnar deviation. Each participant will perform two trials with each hand, with a 30-second rest between trials. The highest score obtained from the dominant hand will be recorded for analysis.
General Health Survey-12 | 8 weeks
  A self-report tool developed by David Goldberg to screen individuals' mental health and determine their overall psychological health level. It is used to identify conditions such as depression, anxiety, impaired social functioning, and psychological stress at an early stage. It was developed to identify individuals at risk of mental health issues in non-clinical populations and is frequently used in community screenings, primary care settings, and epidemiological studies.
Cognitive Reserve Index Questionnaire | 8 weeks
  Nucci et al. developed and standardized the Cognitive Reserve Index Questionnaire to measure an individual's cognitive reserve in three dimensions: education, work activity, and participation in leisure activities. This questionnaire is applied among items by taking into account the frequency of an individual's participation in cognitively challenging activities throughout their life. The validity and reliability of the questionnaire for the Turkish population were established by Özakbaş et al. in 2021.It's a questionnaire that collects information under three main headings. Scores from all three domains are normalized and combined to calculate an overall cognitive reserve score. Low scores indicate low cognitive reserve, while high scores indicate high cognitive reserve.
Body mass index | 8 weeks
  Body mass index is calculated by dividing body weight by the square of height in meters (kg/m2).
Waist/Height Ratio | 8 weeks
  Waist circumference is measured in centimeters at the narrowest part of the waist, at the level of the lowest rib at the end of exhalation, over underwear while the individual is standing, using a loose, non-stretchable tape measure. Height is also measured in centimeters, and waist circumference is divided by height, calculating the waist-to-height ratio.
Waist-hip ratio | 8 weeks
  Waist-hip ratio will be determined by dividing waist circumference (cm) by hip circumference (cm) and recorded in centimeters.

IPD SHARING:
Plan to Share IPD: No